CLINICAL TRIAL: NCT02837770
Title: Analgesic Effect of Topical and Oral Diclofenac on Pain Related to Intravitreal Injections, a Randomized, Triple-arm, Double-blind, Placebo-controlled Study.
Brief Title: Effect of Topical and Oral Diclofenac on Pain Related to Intravitreal Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Constantinos D. Georgakopoulos, MD, PhD, Associate Professor of Ophthalmology, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 72/2016
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-10

CONDITIONS: Pain
Keywords: pain; intravitreal injection; anti-VEGF; diclofenac eye drops; oral diclofenac; Short Form of McGill Pain Questionnaire
MeSH Terms: conditions — Pain | interventions — Diclofenac; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pacebo pill and Diclofenac Eye Drops (Active Comparator): Pacebo pill will be administered 4 hours before the IVI and one drop of Diclofenac 0.1% will be instilled 45' prior to the IVI.
  Interventions: Drug: Diclofenac Eye Drops; Drug: Pacebo pill
- Oral Diclofenac and Diclofenac Eye Drops (Active Comparator): One Diclofenac Sodium sustained-release 75mg tablet administered per os 4 hours prior to the IVI and one drop of Diclofenac 0.1% will be instilled 45' prior to the IVI.
  Interventions: Drug: Oral Diclofenac; Drug: Diclofenac Eye Drops
- Pacebo pill and Artificial Tears (Placebo Comparator): Pacebo pill will be administered 4 hours before the IVI and one drop Artificial Tears will be instilled 45' prior to the IVI.
  Interventions: Drug: Pacebo pill; Drug: Artificial Tears

INTERVENTIONS:
Drug: Diclofenac Eye Drops — One drop of Diclofenac 0.1% will be instilled 45' prior to the IVI.
  Other Names: DENACLOF EY.DRO.SOL 0.1% (W/V)
  Arms: Pacebo pill and Diclofenac Eye Drops
Drug: Pacebo pill — Pacebo pill will be administered 4 hours before the IVI.
  Arms: Pacebo pill and Diclofenac Eye Drops
Drug: Oral Diclofenac — One Diclofenac Sodium sustained-release 75mg tablet administered per os 4 hours prior to the IVI.
  Other Names: VOLTAREN S.R.F.C. 75MG/TAB
  Arms: Oral Diclofenac and Diclofenac Eye Drops
Drug: Diclofenac Eye Drops — One drop of Diclofenac 0.1% will be instilled 45' prior to the IVI.
  Other Names: DENACLOF EY.DRO.SOL 0.1% (W/V)
  Arms: Oral Diclofenac and Diclofenac Eye Drops
Drug: Pacebo pill — Pacebo pill will be administered 4 hours before the IVI.
  Arms: Pacebo pill and Artificial Tears
Drug: Artificial Tears — One drop Artificial Tears will be instilled 45' prior to the IVI.
  Other Names: TEARS NATURALE 0,1%+0,3% EY.DRO.SOL.
  Arms: Pacebo pill and Artificial Tears

SUMMARY:
The analgestic efffect of Diclofenac Sodium 0.1% Eye Drops and a combination of Diclofenac Sodium 0.1% Eye Drops and oral Diclofenac Sodium sustained-release 75mg tablets on pain related to intravitreal injections will be evalutated.

Pain perception will be assessed by the Short Form of the McGill Pain Questionnaire.

DETAILED DESCRIPTION:
Intravitreal injection (IVI) is a preferred route of administration of drugs in the posterior segment of the eye. Intravitreal injection of anti-VEGFs constitutes the mainstay for the treatment of various retinal diseases such as AMD, RVO, DME etc.

The procedure of the IVI is, however, associated with a level of discomfort for the patient.

Nonsteroidal anti-inflammatory drugs (NSAIDs) inhibit the activity of cyclooxygenase-1 and cyclooxygenase-2, and thereby, the synthesis of prostaglandins and thromboxanes. Cyclooxygenase-2 inhibition leads to the anti-inflammatory, analgesic and antipyretic effects of NSAIDs.

Ophthalmic NSAIDs constitute an established and effective treatment option for the management of inflammation and pain associated with cataract surgery and of pain associated with corneal refractive surgery, for inhibition of intraoperative miosis and for the treatment of seasonal allergic conjunctivitis.

The primary goal of this study is to assess the analgesic effect of DIclofenac 0.1% Eye Drops a topical NSAID, as well as a combination of Diclofenac 0.1% Eye Drops and oral Diclofenac Sodium sustained-release (SR) 75mg tablets on pain related to intravitreal injections immediately after and up to six hours post-IVI.

A number of patients scheduled to undergo IVIs of anti-VEGFs will be randomized and divided in three groups. All patients must have already undergone at least one IVI. In patients receiving IVIs in both eyes only one eye will be included in the study.

The patients of the first group will receive placebo pill 4 hours before the IVI and Diclofenac 0.1 % Eye Drops 45 minutes prior to the injection.

The patients of the second group will recieve oral Diclofenac Sodium SR 75mg/tb 4 hours prior to the injection and Diclofenac 0.1% Eye Drops 45 minutes prior to the injection.

The patients of the third group will receive placebo pill 4 hours and Artificial Tears 45 minutes prior to the injection.

Patients will be required to complete the greek version of the short form McGill Pain Questionnaire (SF-MPQ) comprising of the Visual Analogue Scale, the main component of the SF-MPQ and the Present Pain Intensity Scale immediately after the injection and 6 hours post-IVI.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be patients of the Medical Retina Department of our Clinic, who are scheduled to receive IVIs of ranibizumab (Lucentis; Novartis Pharma S.A.S., Huningue, France) or aflibercept (Eylea; Bayer Healthcare Pharmaceuticals, Berlin, Germany) in one eye and had already undergone at least one IVI of an anti-VEGF agent.

Exclusion Criteria:

* History of previous eye surgery other than cataract extraction surgery, herpetic eye disease, uncontrolled glaucoma, uveitis, active conjunctivitis, keratitis and bullous keratopathy, a previously known allergic response to diclofenac or other NSAIDs and salicylates, any contraindication to NSAIDs administration such as cardiovascular disease, gastrointenstinal disease with risk of GI ulceration,bleeding and perforation, renal and hepatic disease and any systemic or topical use of NSAIDs or any use of sedative medications within 7 days from the visit and during the day of IVI.
* Patients with poor cooperation in understanding and answering the questions of the SF-MPQ, including the visual analogue scale (VAS).
* Unsuccessful blinding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Assessment of topical and oral Diclofenac's analgesic effect in patients undergoing intravitreal injections of anti-VEGFs as measured by the Visual Analogue Scale. | Immediately after injection

SECONDARY OUTCOMES:
Assessment of topical and oral Diclofenac's analgesic effect in patients undergoing intravitreal injections of anti-VEGFs as measured by the Visual Analogue Scale. | Six hours after injection
Assessment of oral and topical Diclofenac's analgesic effect after intravitreal injections of anti-VEGFs as measured by the Main Component of the Short Form of the McGill Pain Questionnaire | Immediately after injection
Assessment of oral and topical Diclofenac's analgesic effect after intravitreal injections of anti-VEGFs as measured by the Main Component of the Short Form of the McGill Pain Questionnaire | Six hours after injection
Assessment of oral and topical Diclofenac's analgesic effect after intravitreal injections of anti-VEGFs as measured by the Present Pain Intensity score | Immediately after injection
Assessment of oral and topical Diclofenac's analgesic effect after intravitreal injections of anti-VEGFs as measured by the Present Pain Intensity score | Six hours after injection

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Georgakopoulos, MD, Phd, Principal Investigator — Associate Professor of Ophthalmology, Medical School, University of Patras, Greece
Locations (1):
- University Hospital of Patras, Pátrai, Achaea, Greece

IPD SHARING:
Plan to Share IPD: Undecided